CLINICAL TRIAL: NCT02594891
Title: Effect of 8.5 F Plastic Stent Without Proximal Flap on Prevention of Post-ERCP Cholangitis on Patients With choledocholithiasis--a Prospective Randomized Trial
Brief Title: Effect of 8.5 F Plastic Stent Without Proximal Flap on Prevention of Post-ERCP Cholangitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: First People's Hospital of Hangzhou (Other)
Responsible Party: Principal Investigator, Jianfeng Yang, Deputy irector, First People's Hospital of Hangzhou
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2011-001-004
Record Dates: First submitted 2015-11-01; First posted 2015-11-03 (Estimated); Last update posted 2016-05-24 (Estimated); Status verified 2016-05

CONDITIONS: Cholangitis; Complication
Keywords: cholangitis; endoscopic retrograde cholangiopancreatography; complication
MeSH Terms: conditions — Cholangitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- endoscopic retrograde biliary drainage (Experimental): Patients will undergo endoscopic retrograde biliary drainage (ERBD) with 8.5 F plastic stent with proximal flap when bile duct stones were removed clearly with ERCP. The stent will be taken out with endoscopy three months later if not discharge self-driven.
  Interventions: Device: endoscopic retrograde biliary drainage
- endoscopic nasobiliary drainage (Placebo Comparator): Patients will undergo endoscopic nasobiliary drainage (ENBD) when bile duct stones were removed clearly with ERCP. The nose bile duct will be pulled out 3-5 days later if no cholangitis occurrence.
  Interventions: Device: endoscopic nasobiliary drainage

INTERVENTIONS:
Device: endoscopic retrograde biliary drainage — A 8.5 F plastic stent with proximal flap （XinChang medical instrument co., LTD,Shanghai, China) will be inserted into common bile duct with standard procedure.
  Arms: endoscopic retrograde biliary drainage
Device: endoscopic nasobiliary drainage — A nose bile duct（XinChang medical instrument co., LTD,Shanghai, China) will be inserted into common bile duct with standard procedure.
  Arms: endoscopic nasobiliary drainage

SUMMARY:
Cholangitis is one of the main complications of endoscopic retrograde cholangiopancreatography (ERCP). Plastic biliary stent was used to prevent the occurrence of post-ERCP cholangitis, but the stent should be taken out 1-2 weeks after ERCP with endoscope again. 8.5 F plastic stent with proximal flap can discharge self-driven from biliary to the gut, it has the advantage of avoiding pulling stent out with endoscope again. The purpose of this study is to explore 8.5 F plastic stent with proximal flap on preventing post-ERCP cholangitis of ERCP in patients with choledocholithiasis.

DETAILED DESCRIPTION:
Since its introduction in 1968, endoscopic retrograde cholangiopancreatography (ERCP) has become a commonly performed endoscopic procedure, and the first choice in the management of choledocholithiasis. Although as an endoscopic minimally invasive procedure, there are still certain complications of ERCP, cholangitis is one of the main complications. In European and American countries, plastic biliary stent was used to prevent the occurrence of post-ERCP cholangitis, but the stent should be taken out 1-2 weeks after ERCP with endoscope again. In China endoscopic nasobiliary drainage is usually adopted to prevent post-ERCP cholangitis. Although nose bile duct was more convenient to pull out without endoscope again, but patients often feel nose pharynx ministry unwell obviously. 8.5 F plastic stent with proximal flap can discharge self-driven from biliary to the gut, it has the advantage of avoiding pulling stent out with endoscope again. The purpose of this study is to explore 8.5 F plastic stent with proximal flap on preventing post-ERCP cholangitis of ERCP in patients with choledocholithiasis.

ELIGIBILITY:
Inclusion Criteria:

Obtention of a written informed consent; Patient with choledocholithiasis; Common bile duct stones are removed clearlly.

Exclusion Criteria:

No written informed consent; Combined with acute pancreatitis, acute cholangitis pre-ERCP; Patient under 18 or over 75 years.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2015-11; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Post-ERCP cholangitis | three months
  The rate and severity of post-ERCP cholangitis will compared between two groups.

SECONDARY OUTCOMES:
adverse events | three months
  Number of participants with adverse events; type, frequency and intensity of adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaofeng Zhang, M.S, Study Director — First People's Hospital of Hangzhou
Locations (1):
- Hangzhou First People's Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] ASGE Standards of Practice Committee; Anderson MA, Fisher L, Jain R, Evans JA, Appalaneni V, Ben-Menachem T, Cash BD, Decker GA, Early DS, Fanelli RD, Fisher DA, Fukami N, Hwang JH, Ikenberry SO, Jue TL, Khan KM, Krinsky ML, Malpas PM, Maple JT, Sharaf RN, Shergill AK, Dominitz JA. Complications of ERCP. Gastrointest Endosc. 2012 Mar;75(3):467-73. doi: 10.1016/j.gie.2011.07.010. No abstract available. PMID 22341094